CLINICAL TRIAL: NCT07143864
Title: Efficacy and Safety of Stapokibart for Primary Cutaneous Amyloidosis: A Randomized, Double-blind, Placebo-controlled Study
Brief Title: Efficacy and Safety of Stapokibart for Primary Cutaneous Amyloidosis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital of Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Aijun Chen, Department of Dermatology, The First Affiliated Hospital of Chongqing Medical University, First Affiliated Hospital of Chongqing Medical University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CQMU-2025-215
Record Dates: First submitted 2025-08-13; First posted 2025-08-27 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Primary Cutaneous Amyloidosis
Keywords: primary cutaneous amyloidosis; Stapokibart
MeSH Terms: conditions — Amyloidosis, Primary Cutaneous

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Stapokibart (Experimental)
  Interventions: Biological: Stapokibart
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo drug

INTERVENTIONS:
Biological: Stapokibart — A humanized monoclonal antibody that targets the interleukin (IL)-4 receptor subunit alpha
  Arms: Stapokibart
Other: Placebo drug — Placebo drugs without Stapokibart
  Arms: Placebo

SUMMARY:
This trial is planned to investigate the efficacy and safety of Stapokibart (an IL-4 receptor antagonist) in patients with PCA.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females aged 18 to 75 years, with a diagnosis of PCA confirmed by skin biopsy, and an IGA score of ≥3, a AASI score of ≥5, and a BSA involvement of ≥5%.
2. Subjects who have received at least 4 weeks of mid-to-high potency or at least 2 weeks of very high potency topical corticosteroids (TCS) or an adequate course of systemic corticosteroids within the 6 months prior to screening, but with an inadequate response; or subjects who are unable to receive the above treatments due to adverse reactions or potential risks.
3. Prior to the first dose, subjects must have used a moisturizer continuously for at least 1 week, once daily, and must continue to use it throughout the study period.
4. Able to understand and complete study-related questionnaires.
5. Able to read, understand, and are willing to sign the informed consent form.
6. Willing and able to comply with study visits and related procedures.
7. Women of childbearing potential must agree to use contraception (such as intrauterine devices, oral contraceptives, or condoms) during the study and for 6 months after the study ends; must have a negative serum pregnancy test within 7 days before the first dose and must not be breastfeeding; male subjects must agree to use contraception during the study and for 6 months after the study ends.

Exclusion Criteria:

1. Use of any of the following treatments within 4 weeks prior to randomization: a. Immunosuppressants or immunomodulators, such as systemic corticosteroids, cyclosporine, mycophenolate mofetil, interferon gamma (IFN-γ), azathioprine, methotrexate, and Janus kinase (JAK) inhibitors; b. UV phototherapy; c. Systemic traditional Chinese medicine (TCM) treatment.
2. Use of topical corticosteroids (TCS), topical calcineurin inhibitors (TCI), TCM, or phosphodiesterase 4 (PDE-4) inhibitors within 2 weeks prior to randomization.
3. Receipt of anti-IL-4R monoclonal antibodies, anti-IgE monoclonal antibodies, or other biologics within 12 weeks or 5 half-lives (whichever is longer) prior to randomization.
4. Receipt of live attenuated vaccines within 12 weeks prior to randomization or planned vaccination during the study period.
5. Use of antihistamines within 1 week prior to randomization (subjects who have been on a stable dose of antihistamines for at least 7 days prior to randomization and plan to continue during the study period may be included).
6. Receipt of allergen-specific immunotherapy (desensitization therapy) within 6 months prior to randomization.
7. Presence of any skin comorbidities that may interfere with study assessments, including but not limited to scabies, cutaneous T-cell lymphoma, psoriasis, etc.
8. Previous receipt of at least 12 consecutive doses of anti-IL-4Rα or IL-13 monoclonal antibodies with inadequate clinical response (defined as failure to achieve AASI 50 during treatment).
9. Presence of any other significant medical history that the investigator deems would pose a risk to the subject's safety or be poorly controlled if the subject participates in the study, in addition to PCA.
10. History of known or suspected immunosuppression (immunodeficiency), including a history of invasive opportunistic infections (such as histoplasmosis, listeriosis, coccidioidomycosis, pneumocystosis, and aspergillosis), even if the infection has resolved; or unusual frequency, recurrence, or chronicity of infections (at the investigator's discretion).
11. Subjects with any type of active malignancy or a history of malignancy (except for cervical cancer that has been cured for more than 5 years prior to the screening period, or non-metastatic squamous cell carcinoma of the skin, basal cell carcinoma, and papillary thyroid cancer).
12. Presence of active Mycobacterium tuberculosis infection.
13. Subjects with severe liver or kidney function impairment during the screening period, such as aspartate aminotransferase or alanine aminotransferase >2 times the upper limit of normal (ULN), total bilirubin >1.5 times ULN, serum creatinine >1.2 times ULN, etc.
14. Presence of active hepatitis during the screening period, or positive for hepatitis B surface antigen (HBsAg), or positive for hepatitis B core antibody (HBcAb) and HBV-DNA, or positive for hepatitis C virus (HCV) antibody and HCV-RNA.
15. Positive for HIV antibody during the screening period, or history of HIV infection.
16. Positive for Treponema pallidum antibody during the screening period (subjects who have undergone standard treatment and have a negative non-treponemal antigen serological test may participate in the study).
17. Participation in another clinical trial of a drug or medical device within 12 weeks prior to randomization.
18. Presence of chronic active or acute infection requiring systemic treatment with antibiotics, antivirals, antiparasitics, antiprotozoals, or antifungals within 4 weeks prior to randomization. After resolution of the infection, the subject may be re-screened once.
19. Subjects who plan to undergo major surgical procedures during the study period.
20. Pregnant or breastfeeding women.
21. Subjects with a history of alcoholism, drug abuse, or known drug dependence.
22. History of atopic keratoconjunctivitis involving the cornea.
23. Any medical or psychiatric conditions that the investigator deems would pose a risk to the subject, interfere with participation in the study, or confound the interpretation of study results.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The percentage of subjects achieving AASI-75 at Week 16 of treatment | At the end of treatment at 16 weeks
  AASI: Amyloidosis Area and Severity Index. The minimum and maximum values: 0-72. Higher scores mean more serious situations.
  AASI-75: A 75% or greater improvement from baseline in the AASI. The minimum and maximum values: 0%-100%. Higher scores mean a better outcome.

SECONDARY OUTCOMES:
The percentage of subjects with a weekly average reduction of≥4 points in PP-NRS score at Week 16 of treatment compared to baseline | At the end of treatment at 16 weeks
  PP-NRS: Peak Pruritus Numerical Rating Scale. The minimum and maximum values: 0-10. Higher scores mean more serious situations.
The percentage of subjects with an IGA score of 0 or 1 and a reduction of≥2 points compared to baseline. | At the end of treatment at 16 weeks
  IGA: Investigator Global Assessment. The minimum and maximum values: 0-4. Higher scores mean more serious situations.
The percentage of subjects achieving AASI-50 compared to baseline. | At the end of treatment at 16 weeks
  AASI: Amyloidosis Area and Severity Index. The minimum and maximum values: 0-72. Higher scores mean more serious situations.
  AASI-50: A 50% or greater improvement from baseline in the AASI. The minimum and maximum values: 0%-100%. Higher scores mean a better outcome.
The percentage of subjects with a weekly average reduction of≥3 points in PP-NRS score compared to baseline | At the end of treatment at 16 weeks
  PP-NRS: Peak Pruritus Numerical Rating Scale. The minimum and maximum values: 0-10. Higher scores mean more serious situations.
Change rates in BSA involvement compared to baseline. | At the end of treatment at 16 weeks
  BSA: Body Surface Area. The minimum and maximum values: 0-100%. Higher scores mean more serious situations.
Changes in DLQI scores compared to baseline. | At the end of treatment at 16 weeks
  DLQI: Dermatology Life Quality Index. The minimum and maximum values: 0-30. Higher scores mean more serious situations.
Changes in absolute eosinophil counts in complete blood counts compared to baseline. | At the end of treatment at 16 weeks
Changes in IgE levels in complete blood counts compared to baseline. | At the end of treatment at 16 weeks
Changes in histopathology of skin lesions compared to baseline in some subjects | At the end of follow-up at 28 weeks

OTHER OUTCOMES:
Safety Endpoints:Including the occurrence of AEs(Adverse Events),and abnormalities in laboratory tests,physical examinations,and vital signs. | At the end of treatment at 16 weeks

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-06-04): https://cdn.clinicaltrials.gov/large-docs/64/NCT07143864/Prot_SAP_000.pdf
  • Informed Consent Form (2025-03-31): https://cdn.clinicaltrials.gov/large-docs/64/NCT07143864/ICF_001.pdf